CLINICAL TRIAL: NCT01110603
Title: A Phase Ib Dose Escalation Study of MK-4827 in Combination With Carboplatin, Carboplatin/Paclitaxel and Carboplatin/Liposomal Doxorubicin in Patients With Advanced Solid Tumors
Brief Title: A Study of MK-4827 in Combination With Standard Chemotherapy in Participants With Advanced Solid Tumors (MK-4827-008 AM1)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010_528; MK-4827-008
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2012-03

CONDITIONS: Cancer: Solid Tumors
Keywords: Cancer; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — niraparib; Carboplatin; Paclitaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MK-4827 + carboplatin (Experimental)
  Interventions: Drug: MK-4827; Drug: carboplatin
- MK-4827 + carboplatin/paclitaxel (Experimental)
  Interventions: Drug: MK-4827; Drug: carboplatin; Drug: paclitaxel
- MK-4827 + carboplatin/liposomal doxorubicin (Experimental)
  Interventions: Drug: MK-4827; Drug: carboplatin; Drug: liposomal doxorubicin

INTERVENTIONS:
Drug: MK-4827 — Capsules, orally, once daily, on Days 1 and 3 of each 21- or 28-day Cycle, at the assigned dose level, starting at 40 mg per dose.
Drug: carboplatin — Intravenous infusion, at AUC 5, once, on Day 3 of each 21- or 28-day cycle
Drug: paclitaxel — Intravenous infusion, 175 mg/m2, once, on Day 3 of each 21-day cycle
  Arms: MK-4827 + carboplatin/paclitaxel
Drug: liposomal doxorubicin — Intravenous infusion, 30 mg/m2, once, on Day 3 of each 28-day cycle
  Arms: MK-4827 + carboplatin/liposomal doxorubicin

SUMMARY:
This study will find the dose limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended Phase 2 dose (RPTD) of MK4827 when administered in combination with standard doses of carboplatin, or carboplatin/paclitaxel, or carboplatin/liposomal doxorubicin in the treatment of advanced solid cancers in adults.

DETAILED DESCRIPTION:
The decision to discontinue new enrollment is not related to any concerns about the safety profile of the product.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a locally advanced or metastatic solid tumor for which carboplatin, carboplatin/paclitaxel, or carboplatin/liposomal doxorubicin are the standard of care.
* Participant has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.

Exclusion Criteria:

* Participant has had chemotherapy, radiotherapy, or biological therapy within 4 weeks prior to entering the study.
* Participant has had more than two prior lines of chemotherapy.
* Participant has known central nervous system metastases or a primary central nervous system tumor.
* Participant is pregnant or breastfeeding or expecting to conceive during the timeframe of the study.
* Participant is known to be human immunodeficiency virus (HIV) positive.
* Participant has a history of Hepatitis B or C.
* Participant has a symptomatic pleural effusion.
* Participant with a left ventricular ejection fraction (LVEF) below the institutional norm, or with prior exposure to doxorubicin is not eligible for the MK4827 + carboplatin/liposomal doxorubicin study arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | Each cycle (21 or 28 Days)

SECONDARY OUTCOMES:
Number of participants with clinical and laboratory adverse events (AEs) | Baseline to 30 days post last dose